CLINICAL TRIAL: NCT01114802
Title: Project Onward: an Innovative E-health Intervention for Cancer Survivors
Brief Title: E-health Intervention for Cancer Survivors
Acronym: Onward
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Mohr, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00026896
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2013-06

CONDITIONS: Cancer
Keywords: Cancer survivors; Anxiety; Depression; Technology Assisted; Internet
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Project Onward website + social network (Experimental): This arm has the website which includes 8 weeks of Internet-based cognitive behavioral therapy combined with discussion and support from a group of up to 8 other cancer survivors.
  Interventions: Behavioral: Project Onward website + social network
- Project Onward website (Active Comparator): This arm has the website which includes 8 weeks of Internet-based cognitive behavioral therapy.
  Interventions: Behavioral: Project Onward website

INTERVENTIONS:
Behavioral: Project Onward website + social network — The website will include 8 weeks of Internet-based cognitive behavioral therapy combined with discussion and support from a group of up to 8 other cancer survivors.
  Arms: Project Onward website + social network
Behavioral: Project Onward website — Access to an interactive website that provides 8 weeks of Internet-based cognitive behavioral therapy.
  Arms: Project Onward website

SUMMARY:
This study will develop and examine the effectiveness of an intervention that utilizes multiple telecommunications technologies to improve cancer survivors' access to mental health care and increase their ability to manage the high risk transition time from active cancer treatment to survivorship. The intervention, referred to as Project Onward, uses an interactive website, e-mail, telephone, and an online social network. The purpose of this study is to pilot a novel intervention that can reduce costs, examine methods to improve adherence to internet based treatment and overcome numerous barriers to treatment for mental health concerns.

DETAILED DESCRIPTION:
Nearly 65% of those with cancer diagnoses will survive for at least 5 years, with approximately 10.5 million cancer survivors in the United States. The time of transition for cancer patients, from active treatment to survivorship, has been identified as a time of high risk for depression and anxiety. Cancer survivors experience higher rates of anxiety and depression than those without a cancer history. Research has identified fear of recurrence, perceived loss of support, and social pressure to resume a "normal" life, among other phenomena, as sources for this emotional distress. However, only about 20% of all patients referred for psychotherapy ever enter treatment and of those who initiate treatment, nearly half drop out before completion. This suggests that there are significant barriers to receiving care. These barriers may be even higher for cancer survivors struggling with issues related to re-entry, such as returning to work, resuming household responsibilities and managing residual symptoms such as fatigue or pain.

The internet promises to provide inexpensive access to treatment at any time of the day or night. Unfortunately, the potential for internet delivered services has not been realized. Studies examining treatments that simply provide access to an internet site commonly result in very high dropout after the first site visit, and typically little or no improvement target symptoms. A variety of methods to improve responses to internet interventions have been examined. In general, e-mail support improves adherence and telephone support can improve adherence even more. Another type of support that has only begun to be investigated is the use of social networks to help maintain adherence.

This intervention will combine a variety of outreach methods, including telephone, email and an online social network, to increase adherence and promote the use of the website and the skills it teaches.

ELIGIBILITY:
Inclusion Criteria:

1. Any cancer diagnosis
2. Has completed treatment for cancer and is currently in full remission.
3. ECOG performance Status of < 3.
4. No history of hospitalization for psychiatric reasons with in the past 5 years.
5. Has a telephone, e-mail account, computer, and broadband access to the Internet.
6. Has familiarity with using the Internet that allows for adequate navigation of website.
7. Is able to speak and read English.
8. Is at least 19 years of age.
9. Is able to give informed consent.

Exclusion Criteria:

1. Has hearing or voice impairment that would prevent participation in assessments or coach treatment arm
2. Has visual impairment that would prevent use of the website and completion of assessment materials.
3. Diagnosis of basal or squamous cell skin cancers

3) Has physical impairments that would limit use of the computer. 4) Meets criteria for dementia by scoring < 25 on the Telephone Interview for Cognitive Status (TICS).

5) Is diagnosed with a psychotic disorder, bipolar disorder, dissociative disorder, current post-traumatic stress disorder (PTSD), current substance abuse, or other diagnosis for which participation in a clinical trial of an internet intervention may be either inappropriate or dangerous, or has been hospitalized for psychiatric reasons within the past 5 years. Patients with substance abuse diagnoses who have been abstinent for 3 months will be admitted if otherwise eligible.

6) Is currently receiving individual psychotherapy or planning to receive psychotherapy during the 8-week treatment phase of the study.

7) Is planning to be out of town or unavailable for treatment for 2 weeks or more during the scheduled treatment time.

8) Exhibits severe suicidality, including ideation, plan, and intent. 9) Has initiated treatment with an antidepressant in past 10 days. Once patients have been on a stable dose for 10 days and do not have an appointment with a physician or psychiatrist to change this dose, the patient will be eligible based on this criterion.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Depression, as measured by the Hospital Anxiety and Depression Scale (HADS) | Measured at baseline, 4 weeks, 8 weeks and 12 weeks

SECONDARY OUTCOMES:
Website utilization (e.g., number of logins, average visit length, total time spent on the site, number of exercises completed) | From baseline through 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David C. Mohr, Ph.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States